CLINICAL TRIAL: NCT00515242
Title: Therapeutic Massage for Generalized Anxiety Disorder
Acronym: CALM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21AT002560 (NIH); R21AT002560 (NIH)
Record Dates: First submitted 2007-08-09; First posted 2007-08-13 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Generalized Anxiety Disorder
Keywords: massage therapy; relaxation treatments
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Massage; Hyperthermia, Induced

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Therapeutic massage
  Interventions: Behavioral: massage
- 2 (Active Comparator): Thermotherapy
  Interventions: Behavioral: thermotherapy
- 3 (Placebo Comparator): Relaxation
  Interventions: Behavioral: relaxing environment

INTERVENTIONS:
Behavioral: massage — therapeutic massage
  Arms: 1
Behavioral: thermotherapy — heat therapy
  Arms: 2
Behavioral: relaxing environment — time in a relaxing environment
  Arms: 3

SUMMARY:
The purpose of this study is to compare the relative effectiveness of three relaxation treatments (therapeutic massage, thermotherapy, and time in a relaxing environment) in reducing anxiety in persons with Generalized Anxiety Disorder.

DETAILED DESCRIPTION:
Anxiety and stress are costly problems that afflict millions of American adults. Together, they are among the most common reasons for which adults use complementary and alternative medical (CAM) therapies as well as more conventional relaxation therapies. Although massage is one of the most popular CAM treatments for anxiety, its effectiveness for this problem has never been rigorously evaluated. This study is designed to evaluate the effectiveness of massage as a treatment for a diagnosed anxiety disorder. Massage will be compared with two other relaxing treatments: thermotherapy and time in a relaxing environment, which reflect the types of activities that persons with anxiety might try to relieve their symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Member of Group Health, Seattle metropolitan area
* Generalized Anxiety Disorder confirmed by SCID
* At least moderate anxiety

Exclusion Criteria:

* Serious mental health co-morbidity
* Any life threatening condition
* Currently receiving psychotherapy
* Substantial alcohol use
* Contraindications for massage

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2007-09; Primary Completion 2008-10 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
anxiety | 6 months

SECONDARY OUTCOMES:
worry, depression, disability | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen J. Sherman, PhD, MPH, Principal Investigator — Group Health
Locations (1):
- Group Health Research Institute, Seattle, Washington, United States